CLINICAL TRIAL: NCT04967664
Title: An Interventional, Phase III, Double-blind, Randomized, Controlled, Parallel-group, Multi-site, Clinical Trial Evaluating the Efficacy and Safety of Qutenza® in Subjects With Post-surgical Neuropathic Pain
Brief Title: Comparison of Qutenza (8% Capsaicin) With a Low-dose Capsaicin for Treatment of Nerve Pain After Surgery
Acronym: RISE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Averitas Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AV001
Record Dates: First submitted 2021-06-10; First posted 2021-07-19 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Post Surgical Neuropathic Pain
MeSH Terms: interventions — Capsaicin; Drug Delivery Systems

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Qutenza (capsaicin) 8% topical system (Experimental): Qutenza (capsaicin 8% topical system, containing capsaicin 179 mg or capsaicin 640 µg/cm2 of topical system)
  Interventions: Drug: Qutenza (capsaicin) 8% topical system
- Low-dose capsaicin control (Active Comparator): capsaicin 0.04% topical system
  Interventions: Drug: capsaicin 0.04% topical system

INTERVENTIONS:
Drug: Qutenza (capsaicin) 8% topical system — High concentration capsaicin
  Arms: Qutenza (capsaicin) 8% topical system
Drug: capsaicin 0.04% topical system — Low-dose capsaicin control
  Arms: Low-dose capsaicin control

SUMMARY:
This is an interventional, Phase III, double-blind, randomized, controlled, parallel-group, multi-site, clinical trial to confirm the efficacy and safety of repeated topical application of Qutenza (capsaicin 8% topical system) versus low-dose capsaicin control (capsaicin 0.04% topical system) in subjects with moderate to severe postsurgical neuropathic pain (PSNP).

DETAILED DESCRIPTION:
After a Screening Period of up to 19 days, including the Baseline Phase from Day -7 to Day -1, subjects will be allocated to Qutenza or to low-dose capsaicin control topical system (capsaicin 0.04%) at the Randomization Visit. The blinded Treatment Period consists of a Core Phase (Day 1 to Week 12) and an Extension Phase (Week 13 to Week 42), which includes a Follow-up of 14 days

ELIGIBILITY:
Inclusion Criteria:

General

1. The subject has given written informed consent to participate.
2. Female or male subjects aged 18 years or older.
3. For women of childbearing potential: negative pregnancy tests at Screening Visit (Visit 1), the Randomization Visit (Visit 2), and prior to each reapplication of the investigational medicinal product (IMP), and must have agreed to practice medically acceptable methods of birth control.

   Confirmation of diagnosis of chronic moderate to severe PSNP
4. Documented diagnosis of PSNP by the following criteria:

   1. A history of post-surgical pain with a duration of at least 6 months to maximally 60 months that is plausibly related to the surgical intervention as documented on a body map.
   2. Douleur Neuropathique 4 interview (DN4i) of at least 3 out of 7 points at Visit 1.
   3. The pain must extend beyond the scar area to neuroanatomically adjacent skin areas and be related to the site of the surgery.
5. Documented diagnosis of probable or definite PSNP according to the following criteria (Finnerup et al. 2016):

   1. The pain must be associated with sensory signs in the same neuroanatomically plausible distribution. The area of sensory changes may extend beyond, be within, or overlap with the area of pain (criterion for probable neuropathic pain), or
   2. In addition to 5a : Direct surgical evidence (e.g., surgeon´s clear verification of an intraoperative nerve lesion) (criterion for definite neuropathic pain).
6. The subject has moderate to severe pain with a baseline value for 24-hr average pain intensity of at least 4 points on the NPRS. The baseline value is calculated as the average of the 24-hr average pain intensity ratings of the Baseline Phase (Day -7 to Day -1). At least 5 (out of the last 7 days) pain ratings should be available during the Baseline Phase. If less than 5 pain ratings are available in the last 7 days, the subject may be rescheduled for Visit 2 (1 time only) after having received appropriate re-training in the use of the e-diary to ensure compliance.

   Suitability for treatment with IMP
7. The size of the affected painful intact skin area is not larger than the size of 4 standard Qutenza topical systems (1120 cm2).
8. The skin in the area where the IMP will be applied, and that may also contain the scar tissue, is intact, dry, and non-irritated (i.e., there are no signs and symptoms of skin disease, skin irritation, inflammation or injury, such as active herpes zoster lesions, atopic dermatitis, ulceration, wounds). This is reflected by a dermal assessment score of 0 = "no evidence of irritation" or 1 = "minimal erythema, barely perceptible".

   Eligibility with regard to protocol adherence, to allowed pre-treatments and concomitant treatments
9. The subject is willing to adhere to the restricted use of concomitant treatments .
10. The subject experiencing pain is:

    1. currently not receiving treatment for PSNP or
    2. receives a stable systemic treatment for PSNP that started more than 30 days prior to the Randomization Visit (Visit 2).

Non-exhaustive list of examples of types of surgeries with resulting PSNP:

Thoracic surgery Breast surgery Abdominal surgery (cholecystectomy, appendectomy) Donor nephrectomy Gynecologic surgery (hysterectomy, C-section) Varicose vein surgery Inguinal herniotomy Lipoma removal Knee surgery Knee arthroplasty Ankle surgery

Exclusion Criteria:

General or previous treatments

1. The subject received Qutenza before the Randomization Visit (Visit 2) or received a medical device in another clinical trial within 7 days before the Randomization Visit (Visit 2), or

   1. Any former use of topical capsaicin in the area of the PSNP before Visit 2, except for the use of a low-dose (<1%) capsaicin product - but not within 7 days before Visit 2.
   2. The subject participated previously in this clinical trial or participated in another clinical trial for the treatment of PSNP completing less than 3 months ago.
2. A score of 0 out of 5 in all 3 categories of the neurological/sensory examinations, i.e., for warm sensation, pinprick and cold sensation at the Screening Visit (Visit 1).

   Confounding factors
3. The subject reported a 24-hr average pain intensity score of 10 on the NPRS for at least 4 days during the Baseline Phase.
4. Any painful procedure planned during the course of the trial that may, in the opinion of the investigator, affect the efficacy or safety assessments.
5. Subjects with PSNP related to a surgery/condition with a high potential for confounding symptoms, e.g., the pain is at least partially due to pain in deeper structures such as muscles or bones (including referred pain from deeper structures) as listed in examples.
6. Other painful conditions in the body area that is affected by PSNP and may affect efficacy or safety assessments and cannot be discriminated from the target pain by the subject, including infectious, non-infectious, inflammatory or neuropathic conditions which could also be complications related to the previous surgical procedure.

   Non-exhaustive list of examples of types of surgeries/conditions not suitable for eligibility Any surgery performed due to suspected neoplasia: suspected residual neoplasia or metastases Conditions where nociceptive or neuropathic pain has been the reason for the surgery, e.g., failed back surgery, carpal tunnel syndrome or other nerve compression syndromes leading to neuropathic pain, (e.g., meralgia paresthetica) Conditions of projected neuropathic pain (i.e., from inguinal hernia repair) with painful symptoms in the genital region, e.g., the scrotum or vagina Amputations Radicular pain and nerve trunk lesions Scar pain neuroma Complex Regional Pain Syndrome (Type I or Type II)

   Contraindications to IMP
7. Neuropathic pain areas located only on the face, above the hairline of the scalp, and/or in proximity to mucous membranes.
8. Hypersensitivity to capsaicin (i.e., chili peppers or over-the-counter [OTC] capsaicin products), or to any excipients of the IMP or to excipients of the cleansing gel in use and their components, or to topical anesthetics in use and their components.

   Medical history/concurrent condition(s)/other factors
9. Pending litigation due to chronic pain or disability.
10. The subject has a history of alcohol or drug abuse or is actively abusing drugs (including alcohol, medication) during the 1 year prior to the Screening Visit (Visit 1) as judged by the investigator.
11. Evidence or history of severe psychiatric illness/disorder during the 3 years prior to the Screening Visit (Visit 1) that, in the investigator's opinion, may affect efficacy or safety assessments or may compromise the subject's safety during trial participation, e.g., major depression, major anxiety disorder, psychosis, severe personality disorders.
12. Evidence of cognitive impairment including dementia that may interfere with the subject's ability to complete pain assessments requiring recall of the average pain level in the past 24 hrs.
13. Surgical intervention in the last 3 months preceding the Screening Visit (Visit 1) if it is affecting the efficacy or safety assessments, or any scheduled or planned surgery during the trial, with the exception of the Extension Phase if the planned surgery is not expected to affect the efficacy or safety assessments.
14. Patients with current clinically significant disease(s) or condition(s) (including clinically significant cardiovascular disease and/or significant pain in other areas) that may affect efficacy or safety assessments, or any other reason which, in the investigator's opinion, may preclude the subject's participation in the full duration of the trial. Patients with current signs and symptoms consistent with Coronavirus disease 2019 (COVID-19) (e.g., dry cough, dyspnea, sore throat, fatigue, fever) or patients who had those symptoms within the last 14 days prior to screening and had a positive SARS-CoV2 PCR test result.
15. Unstable or poorly controlled blood pressure which, in the opinion of the investigator, would put the subject at risk of severe adverse blood pressure increases upon IMP application.
16. Known or suspected of not being able to comply with the requirements of the trial protocol or the instructions of the trial site staff.
17. Not able to communicate meaningfully with the trial site staff.
18. The subject is an employee of the investigator or trial site, with direct involvement in the proposed trial or other trials under the direction of that investigator or trial site, or is a family member of the employees or the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 409 (Actual)
Dates: Start 2021-07-13 (Actual); Primary Completion 2025-03-07 (Actual); Study Completion 2025-08-28 (Actual)

PRIMARY OUTCOMES:
Change from baseline to the weekly average score of Week 12 in the 24-hr average pain intensity [Core Phase]. | From the Baseline Phase (Day -7 to Day -1) to Visit 6 (Week 12/Day 84).
  For the US. The 24-hr average pain intensity will be assessed and reported in the electronic diary (e-diary) once daily in the evening, using an 11-point numeric pain rating scale (NPRS, from 0 = no pain to 10 = pain as bad as you can imagine).
Change from baseline to the average score of the entire period between Week 2 and Week 12 in the 24-hr average pain intensity [Core Phase]. | From the Baseline Phase (Day -7 to Day -1) to Visit 6 (Week 12/Day 84).
  For non-US countries/regions. The 24-hr average pain intensity will be assessed and reported in the electronic diary (e-diary) once daily in the evening, using an 11-point numeric pain rating scale (NPRS, from 0 = no pain to 10 = pain as bad as you can imagine).

SECONDARY OUTCOMES:
Change from baseline to Week 12 in the treatment area size [Core Phase]. | Visit 2 (Day 1) and at Visit 6 (Week 12/Day 84)
  The treatment area size [cm2] (the treatment area will be comprised of the area identified by the subject as the usually most painful area(s) and/or the area characterized by dynamic mechanical allodynia [DMA] and/or the area of pinprick hyperalgesia) at Visit 2 (Day 1) before investigational medicinal product (IMP) application and at Visit 6 before IMP application (Week 12/Day 84).
Incidence of Treatment-Emergent Adverse Events (TEAEs) [Core Phase] | Visit 2 (Day 1) up to Visit 6 (Week 12/Day 84)
  Documentation of TEAEs (Safety and tolerability) from the start of treatment at Visit 2 (Day 1) up to the end of the Core Phase of the Treatment Period.
Incidence of TEAEs leading to discontinuation [Core Phase] | Visit 2 (Day 1) up to Final Visit (Week 42/Day 294)
  Documentation of TEAEs (Safety and tolerability) from the start of treatment at Visit 2 (Day 1) up to the end of the Core Phase of the Treatment Period.
Change from baseline to the average score of Week 42 in the 24-hr average pain intensity [Extension Phase]. | Baseline Phase (Day -7 to Day -1) up to the Final Visit (Week 42/Day 294).
  The 24-hr average pain intensity will be assessed and reported in the e-diary once daily in the evening, using an 11-point NPRS (from 0 = no pain to 10 = pain as bad as you can imagine).
Change from baseline to Week 42 in the treatment area size [Extension Phase]. | Visit 2 (Day 1) and at Visit 6 (Week 12/Day 84)
  The treatment area size [cm2] (the treatment area will be comprised of the area identified by the subject as the usually most painful area(s) and/or the area characterized by dynamic mechanical allodynia [DMA] and/or the area of pinprick hyperalgesia) at Visit 2 (Day 1) before investigational medicinal product (IMP) application and at Visit 6 before IMP application (Week 12/Day 84).
Change from baseline to the average score of the entire period between Week 2 and Week 42 in the 24-hr average pain intensity [Extension Phase]. | Baseline Phase (Day -7 to Day -1) to Final Visit (Week 42/Day 294).
  The 24-hr average pain intensity will be assessed and reported in the e-diary once daily in the evening using an 11-point NPRS (from 0 = no pain to 10 = pain as bad as you can imagine).
Incidence of TEAEs [Extension Phase] | Visit 2 (Day 1) up to Final Visit (Week 42/Day 294)
  Documentation of TEAEs (Safety and tolerability) from the start of treatment at Visit 2 (Day 1) up to the end of the Core Phase of the Treatment Period.
Incidence of TEAEs leading to discontinuation [Extension Phase] | Visit 2 (Day 1) up to Visit 6 (Week 12/Day 84)
  Documentation of TEAEs (Safety and tolerability) from the start of treatment at Visit 2 (Day 1) up to the end of the Core Phase of the Treatment Period.

CONTACTS AND LOCATIONS:
Locations (64):
- United States (23):
  - Tucson Orthopaedic Institute, Tucson, Arizona
  - ILD Research Center, Vista, California
  - International Spine, Pain, and Performance Center, Washington D.C., District of Columbia
  - South Lake Pain Institute, Clermont, Florida
  - University Clinical Research - DeLand Clinical Research Unit, DeLand, Florida
  - Florida Research Center, Inc., Miami, Florida
  - Clinical Research of West Florida, Tampa, Florida
  - Drug Studies America, Marietta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Neuroscience Research Center, LLC, Overland Park, Kansas
  - Kansas City Bone & Joint Clinic, P.A., Overland Park, Kansas
  - Boston Clinical Trials, Boston, Massachusetts
  - Great Lakes Research Group, Inc., Bay City, Michigan
  - Premier Pain Centers, Shrewsbury, New Jersey
  - Ainsworth Institute of Pain Management, New York, New York
  - Accellacare, Wilmington, North Carolina
  - The Center for Clinical Research, Winston-Salem, North Carolina
  - META Medical Research Institute, LLC, Dayton, Ohio
  - Main Line Spine, King of Prussia, Pennsylvania
  - New Phase Research & Development, Knoxville, Tennessee
  - Expert Pain, Houston, Texas
  - The University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Wasatch Clinical Research, LLC, Salt Lake City, Utah
- France (11):
  - Centre Hospitalier Departemental Vendee - Centre d'evaluation et de Traitement de la Douleur, La Roche-sur-Yon, Pays de la Loire Region
  - CHU de Nantes - Hopital Nord Laennec, Nantes, Pays de la Loire Region
  - CHU Amiens Picardie, Amiens
  - Centre Regional De Lutte Contre Le Cancer (Crlcc) -Centre Paul Papin, Angers
  - Centre Hospitalier Jean Rougier, Cahors
  - Centre Hospitalier Universitaire de Clermont Ferrand, Clermont-Ferrand
  - Centre Hospitalier Regional Universitaire (CHRU) de Lille - Hopital Claude Huriez, Lille
  - Clinique Francois Chenieux, Limoges
  - Cochin Hospital-Paris Descartes University, Paris
  - Groupe Hospitalier Paris saint-Joseph, Paris
  - CHU Poitiers / La Miletrie, Poitiers
- Netherlands (4):
  - VUMC, Amsterdam
  - PT&R, Beek
  - NOCEPTA, Hengelo
  - Leiden University Medical Center (LUMC), Leiden
- Poland (9):
  - Centrum Medyczne Pratia Katowice, Katowice, Silesian Voivodeship
  - Silmedic Sp z o.o. Oddzial w Katowicach, Katowice, Silesian Voivodeship
  - Vitamed Nzoz Im. Edyty Jakubow, Bialystok
  - Nzoz Neuro-Medic, Katowice
  - Linden Centrum Medyczne, Krakow
  - Instytut Zdrowia dr Boczarska-Jedynak, Oświęcim
  - Lubelskie Centrum Diagnostyczne, Świdnik
  - Centrum Badan Medycznych Nigrir, Warsaw
  - FutureMeds sp. z o. o., Wroclaw
- Spain (10):
  - Hospital General Universitario de Alicante, Alicante, Alicante
  - Hospital Universitario de La Princesa, Madrid, Madrid
  - Hospital Clinico Universitario de Valencia, Valencia, Valencia
  - Hospital Del Mar, Barcelona
  - Hospital Universitario de Bellvitge, L'Hospitalet de Llobregat
  - Hospital Universitario La Moraleja, Madrid
  - Hospital Quironsalud Malaga, Málaga
  - Clinica Universidad de Navarra, Pamplona
  - Clinica Gaias, Santiago de Compostela
  - Hospital Clinico Universitario de Valladolid, Valladolid
- United Kingdom (7):
  - Accellacare - (MeDiNova Limited) - Northamptonshire, Corby, Northamptonshire
  - Accellacare - (MeDiNova Limited) - Yorkshire, Shipley, Yorkshire
  - Aberdeen Royal Infirmary (ARI) - NHS Grampian, Aberdeen
  - Accellacare, Coventry
  - Leeds General Infirmary - Leeds Teaching Hospitals NHS Trust, Leeds
  - Accellacare - (MeDiNova Limited) - North London, Northwood
  - MeDiNova South London Quality Research Site, Sidcup